CLINICAL TRIAL: NCT03776955
Title: Beta-blockers or Placebo for Primary Prophylaxis of Oesophageal Varices (BOPPP Trial). A Blinded, Multi-centre, Clinical Effectiveness and Cost-effectiveness Randomised Controlled Trial
Brief Title: Beta-blockers for Oesophageal Varices
Acronym: BOPPP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other); Guy's and St Thomas' NHS Foundation Trust (Other); St George's University Hospitals NHS Foundation Trust (Other); Cardiff University (Other); Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 125861
Record Dates: First submitted 2018-11-30; First posted 2018-12-17 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Cirrhoses, Liver; Oesophageal Varices
MeSH Terms: conditions — Esophageal and Gastric Varices | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo matched control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Carvedilol (Experimental): 6.25 mg or 12.5 mg if tolerated
  Interventions: Drug: Carvedilol
- Oral Placebo (Placebo Comparator)
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — Oral tablet

SUMMARY:
To determine if carvedilol reduces the rate of variceal haemorrhage in patients with cirrhosis and small oesophageal varices

DETAILED DESCRIPTION:
Cirrhosis or liver scarring is an important problem in healthcare in the United Kingdom. 60,000 patients are living with this disease and about 11,000 people every year will die because of it. There are several ways in which patients with this severe form of liver disease become unwell or die and bleeding from the oesophagus or stomach is one. Cirrhosis causes pressure changes inside the abdomen and swelling of veins in the oesophagus (called "varices") which can bleed catastrophically.

The investigators know that when varices are large, treatment can be initiated with medication called beta-blockers to reduce the pressure in the varices. If the varices are small, the medical community is not sure if treatment with beta-blockers will work. This study aims to address this uncertainty.

Patients who are recruited to the study with small varices will be randomised to either beta-blockers or a placebo. Research sites will observe patients closely for 3 years for bleeding from their varices or other complications of cirrhosis or side effects of taking medication. This is the amount of time needed to observe for bleeding when the varices are small. Research sites will review the patients every 6 months including assessing the varices by a camera test called an endoscopy at the beginning and each year until the study is finished.

During the study, patients will be involved with the conduct and management of the research. Patient will also be notified on the trial results at the end of the study. The barriers and facilitators in adjusting the dose of the tablets to optimise treatment effects primary care will be along with patients' views on taking part in the trial, and whether the side effects justify the potential benefits of reducing the risk of bleeding. The investigators estimate this risk could be reduced from 20% of patients having significant bleeding to 10% over 3 years.

The investigators will measure the impact of beta-blockers on the overall costs to the National Health Service (NHS) of caring for people with cirrhosis during the trial, and will also assess the impact of treatment on both mortality and quality of life using a combined measure, the Quality Adjusted Life-Year (QALY). The investigators will use a mathematical prediction model to estimate the impact of treatment on costs, mortality and quality of life over a patient's lifetime and will assess whether any increased costs are justified by better outcomes for patients and represent good value for money for the NHS budget.

Finally, the results of the study will be published in the medical literature and discuss the findings at medical conferences, patient groups and with charities involved in helping patients with cirrhosis such as the British Liver Trust.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Cirrhosis and portal hypertension, defined by any 2 of the following:

   A) Characteristic clinical examination findings; one or more of i) liver function tests ii) haematological panel iii) coagulation profile abnormalities B) Characteristic radiological findings; one or more of i) heterogeneous, small liver with irregular contour ii) splenomegaly iii) ascites iv) varices v) recanalized umbilical vein C) Fibrosis score > stage 4 on liver biopsy D) FibroScan liver stiffness measurement >15 kilo Pascal without other explanation
3. Small oesophageal varices diagnosed within the last 3 months,- defined as <5 mm in diameter or varices which completely disappear on moderate insufflation at gastroscopy.
4. Not received a beta-blocker in the last week
5. Capacity to provide informed consent

Exclusion Criteria:

1. Non-cirrhotic portal hypertension
2. Medium/large oesophageal varices (current or history of), defined as >5 mm in diameter
3. Isolated gastric, duodenal, rectal varices with or without evidence of recent bleeding
4. Previous variceal haemorrhage
5. Red signs accompanying varices at endoscopy
6. Known intolerance to beta blockers
7. Contraindication to beta blocker use i) Heart rate <50 bpm ii) Known 2nd degree or higher heart block iii) Sick sinus syndrome iv) Systolic blood pressure <85 mm Hg v) Chronic airways obstruction (asthma/COPD) vi) Floppy Iris Syndrome vii) CYP2D6 Poor Metaboliser viii) History of cardiogenic shock ix) History of severe hypersensitivity reaction to beta-blockers x) Untreated phaeochromocytoma xi) Severe peripheral vascular disease xii) Prinzmetal angina xiii) New York Heart Association IV heart failure
8. Unable to provide informed consent
9. Child Pugh C cirrhosis
10. Already receiving a beta-blocker for another reason that cannot be discontinued
11. Graft cirrhosis post liver transplantation
12. Evidence of active malignancy without curative therapy planned
13. Pregnant or lactating women
14. Women of child bearing potential not willing to use adequate contraception during the protocol of IMP dosing
15. Patients who have been on a CTIMP within the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Variceal bleeding | 3 years
  Time to first variceal haemorrhage
Health Economic assessment | 3 years
  Assess the cost effectiveness of early intervention with non specific beta blockers in this patient population.

SECONDARY OUTCOMES:
Variceal bleed rate | 1 and 3 years
  Number of variceal bleeds by allocation
Variceal bleeding needing intervention | 3 years
  Number of patients that progress to medium/large varices requiring clinical intervention
Composite of variceal bleed rate and bleeding needing intervention | 3 years
  Composite of variceal bleed rate and bleeding needing intervention. i.e. Unit less measure of rate of ((Number of patients who bled) PLUS (Number of patients who progressed without bleeding)) / (Number of patients in that arm at randomisation) at 3 years ranging from 0 to 1
Clinical decompensation | 3 years
  Number of patients with clinical decompensation (spontaneous bacterial peritonitis, new ascites, new hepatic encephalopathy) in the active and inactive IMP groups
Child Pugh Score for Cirrhosis mortality | 3 years
  Child Pugh Score for Cirrhosis mortalityin the active and inactive IMP groups. Range 5-15. Higher scores represent worse outcomes.
Model for end-stage liver disease (MELD) score | 3 years
  MELD score in the active and inactive IMP groups.Range 6-40. Higher scores represent worse outcomes.
Survival (Overall, liver related, cardio-vascular related) | 3 years
  Survival (Overall, liver related, cardio-vascular related)
Quality of life assessment | 3 years
  Quality of life score using EQ5D-5L in the active and inactive IMP groups. Range 5-25. Higher scores represent worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Mark McPhail, BSc, PhD, MB ChB, Study Director — King's College Hospital NHS Trust; Ben Carter, BSc, PhD, Study Director — King's College London
Locations (4):
- United Kingdom (4):
  - Royal Victoria Hospital, Belfast, Northern Ireland
  - Queen Elizabeth Hospital, Birmingham
  - Royal London Hospital (Barts), London
  - King's College Hosptial NHS Foundation Trust (Denmark Hill), London

IPD SHARING:
Plan to Share IPD: Undecided
To be decided